CLINICAL TRIAL: NCT02985255
Title: Role of Neo-adjuvant Chemotherapy in Organ Preservation in Locally Advanced Squamous Cell Carcinoma of Oral Tongue
Brief Title: Role of Neo-adjuvant Chemotherapy in Tongue Preservation in Locally Advanced Squamous Cell Carcinoma of Oral Tongue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HealthCare Global Enterprise Ltd. (Industry)
Responsible Party: Principal Investigator, Vishal U S Rao, Senior Consultant, HealthCare Global Enterprise Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCG/SX/001/2016
Record Dates: First submitted 2016-09-29; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Tongue Neoplasms; Squamous Cell Carcinoma; Anterior Tongue Squamous Cell Carcinoma
Keywords: Neoadjuvant Chemotherapy; Tongue Malignancy; Squamous Cell Carcinoma
MeSH Terms: conditions — Tongue Neoplasms; Carcinoma, Squamous Cell | interventions — Docetaxel; Cisplatin; Fluorouracil; Radiotherapy; Glossectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Arm (Experimental): Study Subjects, eligible for NACT would undergo a pretreatment workup with Evaluation Under Anesthesia for tumor Mapping and tissue biopsy along with a PET-CT scan. They would undergo 3 cycles of NACT (weekly thrice) with injection Docetaxel, Cisplatin and 5-FU after which reassessment with PET-CT and EUA +/- biopsy would be done. Those achieving CR would undergo adjuvant CTRT while subjects with PR in PET-CT scan will be reclassified based on the biopsy report. If biopsy is negative for malignancy, they will undergo adjuvant CTRT but would undergo surgery if in the PR group. Subjects with SD or PD would undergo surgery. PET-CT and EUA +/- HPE analyses would be repeated on follow-up after 3 months of treatment completion.
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: 5FU; Radiation: Radiotherapy; Procedure: Glossectomy

INTERVENTIONS:
Drug: Docetaxel — Neoadjuvant Arm
Drug: Cisplatin — Neoadjuvant Arm
Drug: 5FU — Neoadjuvant Arm
Radiation: Radiotherapy — Neoadjuvant Arm
Procedure: Glossectomy — Neoadjuvant Arm

SUMMARY:
Patients enrolled for the study, who are eligible for NACT, will undergo a pre-treatment workup comprising of Evaluation Under Anesthesia (EUA) for tumor Mapping and tissue biopsy along with a PET-CT scan. Subsequently, they would undergo 3 cycles of NACT (weekly thrice) with DCF. They would be reassessed with PET-CT and EUA +/- biopsy after the end of the third cycle. Those who are achieving CR would undergo adjuvant CTRT. Subjects who have a PR in the PET-CT scan will be re-classified based on the biopsy report. If they remain in the PR group they will undergo surgery but if the biopsy in is negative for malignancy, they will undergo adjuvant CTRT. Those subjects with SD or PD would undergo surgery. Subsequently, further radiation and/ or chemotherapy will be decided based on the final histopathology (of the surgical specimen) reports.

PET-CT and EUA +/- HPE analyses would be repeated on follow-up after 3 months of treatment completion.

DETAILED DESCRIPTION:
Patients enrolled for the study, who are eligible for Neoadjuvant chemotherapy, will undergo a pre-treatment workup comprising of Evaluation Under Anesthesia (EUA) for tumor Mapping and tissue biopsy along with a PET-CT scan. Subsequently, they would undergo 3 cycles of Neoadjuvant chemotherapy (weekly thrice) with injection Docetaxel, Cisplatin, and 5-FU. They would be reassessed with PET-CT and EUA +/- biopsy after the end of the third cycle. Those who are achieving a Complete Response (CR) would undergo adjuvant chemo-radiotherapy. Subjects who have a partial response (PR) in the PET-CT scan will be re-classified based on the biopsy report. If they remain in the PR group they will undergo surgery. If the biopsy in these patients is negative for malignancy, they will undergo adjuvant chemoradiotherapy. Those subjects with stable disease (SD) or progressive disease (PD) would undergo surgery. Subsequently, further radiation and/ or chemotherapy will be decided based on the final histopathology (of the surgical specimen) reports.

PET-CT and EUA +/- HPE analyses would be repeated on follow-up after 3 months of treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients of newly diagnosed squamous cell carcinoma (well/ moderately/ poorly differentiated) of oral tongue (anterior two third) presenting to Health Care Global Enterprises Ltd between January 2016 to March 2017 will be included in the study.
* Stage III and stage IV (T3, 4 N0-3, M 0) and selected cases of T2 with advanced nodal status will also be included in the study.

Exclusion Criteria:

* Patients having recurrence/ residual disease of oral tongue.
* Patients who have received alternative treatments before being evaluated for NACT
* Patient who are not fit for NACT
* Patient not able to give consent

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Tongue Preservation Rate | At Response evaluation post 3rd CT Cycle (approximately 7 months post recruitment)
  A ratio of the number of study subjects who have achieved a complete response and do not require surgery, after 3 cycles of NaCT to the total number of subjects recruited to the study.

SECONDARY OUTCOMES:
Overall Survival | 2 years post treatment completion
  Overall Survival Rate (Date of diagnosis to date of death or last follow-up) in different sub-cohorts of the study
Progression Free Survival | 2 years post treatment completion
  Progression Free Survival Rate (Primary treatment end date to date of progression or last follow-up) in difference sub-cohorts of the study
Sensitivity and Specificity of PET-CT | At Baseline and after 12-15 weeks (post 3 cycles of NaCT (Typically 3 weeks))
  Ability of PETCT (along with HPE and EUA) to detect response rates in study subjects undergoing NACT for Ca Tongue

CONTACTS AND LOCATIONS:
Overall Officials: Vishal US Rao, MS, Principal Investigator — Dept of Head & Neck Surgery, HealthCare Global Enterprises Ltd.
Locations (1):
- HealthCare Global Enterprises Ltd, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barringer DA, Hutcheson KA, Sturgis EM, Kies MS, Lewin JS. Effect of induction chemotherapy on speech and swallowing function in patients with oral tongue cancer. Head Neck. 2009 May;31(5):611-7. doi: 10.1002/hed.20989. PMID 19107949
- [Background] Kies MS, Boatright DH, Li G, Blumenschein G, El-Naggar AK, Brandon Gunn G, Lewin JS, Steinhaus GD, Sturgis EM. Phase II trial of induction chemotherapy followed by surgery for squamous cell carcinoma of the oral tongue in young adults. Head Neck. 2012 Sep;34(9):1255-62. doi: 10.1002/hed.21906. Epub 2011 Oct 19. PMID 22009800
- [Background] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Background] Blanchard P, Bourhis J, Lacas B, Posner MR, Vermorken JB, Cruz Hernandez JJ, Bourredjem A, Calais G, Paccagnella A, Hitt R, Pignon JP; Meta-Analysis of Chemotherapy in Head and Neck Cancer, Induction Project, Collaborative Group. Taxane-cisplatin-fluorouracil as induction chemotherapy in locally advanced head and neck cancers: an individual patient data meta-analysis of the meta-analysis of chemotherapy in head and neck cancer group. J Clin Oncol. 2013 Aug 10;31(23):2854-60. doi: 10.1200/JCO.2012.47.7802. Epub 2013 Jul 8. PMID 23835714
- [Background] Forastiere AA, Zhang Q, Weber RS, Maor MH, Goepfert H, Pajak TF, Morrison W, Glisson B, Trotti A, Ridge JA, Thorstad W, Wagner H, Ensley JF, Cooper JS. Long-term results of RTOG 91-11: a comparison of three nonsurgical treatment strategies to preserve the larynx in patients with locally advanced larynx cancer. J Clin Oncol. 2013 Mar 1;31(7):845-52. doi: 10.1200/JCO.2012.43.6097. Epub 2012 Nov 26. PMID 23182993